CLINICAL TRIAL: NCT04726488
Title: Periareolar Approach in Minimally Invasive Cardiac Surgery; New Trend.
Brief Title: Periareolar Approach in Minimally Invasive Cardiac Surgery
Acronym: PAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed El Adel Sayed Hassanein Sayed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Periareolar Minimally Invasive
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Periareolar Minimally Invasive Cardiac Surgery

STUDY DESIGN:
Masking Description: All investigators will be blinded (i.e., closed envelop open in the OR to choose which approach will be performed either periareolar Vs infra-mammary approach in minimally invasive cardiac surgery)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periareolar Approach (Experimental): To study the feasibility and safety of "periareolar minimally invasive surgery" protocol in patients undergoing periareolar minimally invasive surgery vs. Control group (inframammary approach).
  Interventions: Procedure: Periareolar Approach in Minimally Invasive Cardiac Surgery (PAMI Technique)
- Inframammary Approach (Active Comparator): To study the feasibility and safety of "periareolar minimally invasive surgery" protocol in patients undergoing periareolar minimally invasive surgery vs. Control group (inframammary approach).
  Interventions: Procedure: inframammary approach

INTERVENTIONS:
Procedure: Periareolar Approach in Minimally Invasive Cardiac Surgery (PAMI Technique) — To study the feasibility and safety of "periareolar minimally invasive surgery" protocol in patients undergoing periareolar minimally invasive surgery vs. Control group (inframammary approach).
  Arms: Periareolar Approach
Procedure: inframammary approach — To study the feasibility and safety of "periareolar minimally invasive surgery" protocol in patients undergoing periareolar minimally invasive surgery vs. Control group (inframammary approach).
  Arms: Inframammary Approach

SUMMARY:
Overall Goal: To study the feasibility and safety of "periareolar minimally invasive surgery" protocol in patients undergoing periareolar minimally invasive surgery vs. Control group (inframammary approach).

* Objective1: Test the hypothesis that, the periareolar approach is more feasible and safer than the inframammary approach.
* Objective2: Identify risk factors that are predictive of the need for periareolar approach.
* Objective3: Assess outcomes and postoperative results of both periareolar and inframammary approach.

DETAILED DESCRIPTION:
The first successful cardiac operation was performed in 1896, in Germany by Rehn (1), followed by the first successful cardiac valve operation in 1912 by Tuffier (2) and the first successful mitral valve operation in 1923 (3).

In 1956, Lillehei repaired multiple valvular lesions through a right thoracotomy using cardiopulmonary bypass (4).

In the 1990s, the success of laparoscopic operations in general surgery renewed an interest in minimally invasive approaches for cardiac surgery. Navia and Cosgrove (5) and Cohn et al. (6) performed the first minimally invasive valve operations via the right parasternal and transsternal approaches. Remarkably, excellent exposure was achieved through smaller incisions, thereby making complex valve repair possible and safe.

In 1996, Carpentier et al. (7) performed the first video-assisted mitral valve repair through a minithoracotomy using ventricular fibrillation. With more experience, video-assisted, 2-dimensional endoscopes and robotics were introduced by Carpentier (7) and Chitwood (8,9).

In 2009 Poffo et al (10,11) describe a new technique of minimally invasive cardiac surgery. He and his colleagues adopting periareolar access for mitral valve surgery since 2006 and published this technique in 2009.

However, due to its feasibility and safety, was soon incorporated as an ideal access for other cardiac pathologies such as tricuspid valve disease, atrial septal defect, atrial fibrillation, and pacemaker leads endocarditis. This led Poffo and his colleagues to publish a long-term result on his technique in 2018 supporting the use of periareolar access as a routine surgical technique for correction of several cardiac pathologies, especially in women. (12)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoes mitral or tricuspid valve surgery.
* lesion of right side of the heart.

Exclusion Criteria:

* patients undergoing aortic valve or CABG surgery.
* surgery of left side of the heart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery | 2 hours
  start from skin incision to cardiopulmonary bypass initiation

SECONDARY OUTCOMES:
rate of surgical site complications | three month
  wound infection, dehiscence, seroma